CLINICAL TRIAL: NCT02975518
Title: Tracking Endothelial Cells in Arterial Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol v 3
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Endothelial Progenitor Cells; Coronary Artery Disease; Vascular Injury; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Vascular System Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intra-venous infusion of Flourodeoxyglucose (Active Comparator): As a control for radio labelled cells, Flourodeoxyglucose will be administered intra-venously at an activity equal to that injected with the labelled endothelial cells.
  Interventions: Biological: Administration of radio labelled endothelial outgrowth cells
- Intra-Arterial infusion of Flourodeoxyglucose (Active Comparator): As a control for radio labelled cells, Flourodeoxyglucose will be administered intra-arterially at an activity equal to that injected with the labelled endothelial cells.
  Interventions: Biological: Administration of radio labelled endothelial outgrowth cells
- Intra-venous injection of radio-labelled endothelial cells (Experimental): Endothelial cells labelled with flourodeoxyglucose will be injected intra-venously with their distribution tracked using PET CT.
  Interventions: Biological: Administration of radio labelled endothelial outgrowth cells
- Intra-Arterial injection of radio-labelled endothelial cells (Experimental): Endothelial cells labelled with flourodeoxyglucose will be injected intra-arterially with their distribution tracked using PET CT.
  Interventions: Biological: Administration of radio labelled endothelial outgrowth cells

INTERVENTIONS:
Biological: Administration of radio labelled endothelial outgrowth cells — Radio labelled endothelial outgrowth cells will be administered to patients undergoing elective coronary angiography and stenting. They will be administered intra-venously and intra-arterially (right radial artery) in separate arms. Migratory behaviour of these cells will be defined using PET CT. Intra-venous and intra-arterial injection of free radio tracer will serve as a control comparator arms.

SUMMARY:
We plan to track the migratory behaviour of culture-expanded enothelial outgrowth cells in the context of vascular injury sustained during elective coronary angiography.

We will use Flouro-deoxyglucose-labelling and PET-CT to track the endothelial cells.

DETAILED DESCRIPTION:
The radial artery is commonly injured following trans-radial cardiac catheterisation and this injury can be demonstrated as a reduction in endothelial function as measured by flow-mediated dilatation which recovers with time (13-15). Thus the radial artery is useful as a model of mechanical arterial injury as radial artery trauma is common and endothelial function can be followed longitudinally with a non-invasive test.

Endothelial progenitor cells localise to sites of arterial injury in animal models both in vitro and in vivo and accelerate re-endothelialisation as well as attenuating neointimal hyperplasia (16-18), This has however not been demonstrated in man.

Our research group, in collaboration with the Scottish Blood Transfusion Service (SNBTS) have developed a good manufacturing practice (GMP)-compliant process for manufacturing an endothelial progenitor cell (EPC) product (SNBTS will manufacture the final product administered to patients). We have also demonstrated in vitro that we can label these cells with the radioisotope 18 F-fluorodeoxyglucose (18F-FDG) and that activity can be detected in as few as 200 cells using a hybrid positron emission and computed tomography (PET-CT) scanner (Biograph mCT Siemens Medical Systems, Erlangen, Germany). We will therefore be able to track the fate of these cells in vivo. The major potential advantage of imaging in this way is that only 18F-FDG associated with EPCs will be delivered to the patient, removing the issue of background attenuation due to "free" circulating 18F-FDG. A similar technique has previously been employed in vivo to track homing of unselected autologous bone marrow cells to infarcted myocardium(19). Following intracoronary delivery using this technique, the authors were able to detect 1.3% - 2.6% of 18F-FDG-labelled cells in the infarcted myocardium. Demonstrating that EPCs are able to home to and integrate at sites of vascular injury in man is a critical step in understanding the role of EPCs in vascular repair

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary angiography for known or suspected ischaemic heart disease

Exclusion Criteria:

1. Previous coronary artery bypass surgery.
2. Planned angiography via the femoral artery as a sole arterial access route
3. Anaemia <10g/L
4. Severe valvular heart disease
5. Acute myocardial infarction within previous three months
6. Cardiac failure (Killip class ≥II).
7. Insulin dependent diabetes mellitus
8. Hepatic failure (Childs-Pugh grades B or C).
9. Renal failure (estimated glomerular filtration rate <25 mL/min).
10. Intercurrent illness including patients with a systemic inflammatory disorder or underlying malignancy.
11. Women of child-bearing age not ensuring reliable methods of contraception.
12. Inability to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Standard uptake value | 0-4 hours
  Standard-uptake values of injured sections of artery will be compared to remote uninjured artery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom